CLINICAL TRIAL: NCT02225145
Title: Fertility Preservation in Females Who Will be Undergoing Gonadotoxic Therapy, Hematopoietic Stem Cell Transplantation, and in Females With Sickle Cell Disease
Brief Title: Fertility Preservation in Women Who Will Have Gonadotoxic Therapy or Hematopoetic Stem Cell Transplantation, and in Women With Sickle Cell Disease
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 140177; 14-CH-0177
Record Dates: First submitted 2014-08-23; First posted 2014-08-26 (Estimated); Last update posted 2018-06-01 (Actual); Status verified 2017-09-20

CONDITIONS: Hemoglobin; Stem Cell Transplant; Aplastic Anemia
Keywords: Bone Marrow Transplant; Fertility; Ovary
MeSH Terms: conditions — Anemia, Aplastic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Background:

- Some treatments for cancer or other diseases can lead to infertility in women. These treatments include chemotherapy, some stem cell transplants, and pelvic radiotherapy. They are called gonadotoxic therapies. Women can now have their eggs frozen before they have these treatments. This may allow them to get pregnant later. Researchers want to learn more about this technology and processes.

Objectives:

- To provide egg freezing for women having gonadotoxic therapies at NIH. To learn more about the effects of these therapies.

Eligibility:

- Women at least 18 years old who are past puberty and before menopause. They must be scheduled to have gonadotoxic therapies.

Design:

* Participants will be screened with medical history and blood and hormone tests. They will also have a physical exam and transvaginal ultrasound.
* Ovary stimulation: participants will have medications injected under the skin. These increase the chance of fertility. This phase will take about 8 20 days. Participants will have blood drawn and transvaginal ultrasound daily or every other day. Some participants will also have blood thinner injected daily.
* Egg retrieval: participants will check in to the hospital. Eggs will be removed with a needle during a short surgery. Participants will be awake but sedated.
* Participants may stay overnight in the hospital.
* They will return every 1 3 days for 1 3 weeks for blood tests.
* Mature eggs will be frozen after egg retrieval and immature eggs (which cannot be fertilized for clinical use) will be used for research. Participants can use their eggs in the future at outside, private fertility clinics to try to become pregnant. If the eggs are stored for more than 5 years, participants must pay for storage.

DETAILED DESCRIPTION:
Treatment with chemotherapeutic drugs, hematopoietic stem cell transplantation, and pelvic radiotherapy for cancer or other serious medical illnesses has the potential to markedly increase the risk of gonadotoxicity leading to infertility in women. Females who are post-menarchal with these risk factors may be candidates for fertility preservation through oocyte cryopreservation before ovarian failure ensues. For example, sickle cell disease (SCD) is the most common hemoglobinopathy in the United States (3). Hypoxic conditions cause the abnormal hemoglobin molecule to undergo sickling which leads to painful microvascular occlusion. SCD is associated with multiple organ system dysfunction as well as neurological and pulmonary complications, which can lead to early mortality. Hematopoietic stem cell transplantation (HSCT) is the only treatment currently available for SCD that results in a complete cure. In patients who have undergone HSCT with a matched sibling, event-free survival has been as high as 85%-95%. Multiple studies have unfortunately demonstrated that infertility and premature ovarian insufficiency are quite common following HSCT. Specifically in our patient population with sickle cell disease, we have recently found largely preserved ovarian function prior to transplantation, but profound gonadotoxicity following transplant (unpublished). This underscores the clinical need for additional, effective fertility preservation methods for our at-risk populations.

ELIGIBILITY:
* INCLUSION CRITERIA:

Subject is able to give consent/assent to participate in the protocol:

* Post-Menarchal females greater than or equal to 7 years old undergoing gonadotoxic therapy, hematopoietic stem cell transplantation, and/or sickle cell disease
* Have a FSH less than or equal to 13 mIU/ml or AMH greater than or equal to 0.5 ng/ml

EXCLUSION CRITERIA:

* Unable to comprehend the investigational nature of the protocol
* Positive pregnancy test
* Ovarian cancer
* Diagnosis of HIV/AIDS

Ages: 7 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2014-08-15; Primary Completion 2016-09-09 (Actual); Study Completion 2017-09-20 (Actual)

PRIMARY OUTCOMES:
Oocyte vitrification | End of Stumulation

CONTACTS AND LOCATIONS:
Overall Officials: Alan H DeCherney, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Practice Committees of the American Society for Reproductive Medicine and the Society for Assisted Reproductive Technology. Mature oocyte cryopreservation: a guideline. Fertil Steril. 2013 Jan;99(1):37-43. doi: 10.1016/j.fertnstert.2012.09.028. Epub 2012 Oct 22. PMID 23083924
- [Background] Practice Committee of American Society for Reproductive Medicine. Fertility preservation in patients undergoing gonadotoxic therapy or gonadectomy: a committee opinion. Fertil Steril. 2013 Nov;100(5):1214-23. doi: 10.1016/j.fertnstert.2013.08.012. Epub 2013 Sep 5. PMID 24011612
- [Background] Dovey S, Krishnamurti L, Sanfilippo J, Gunawardena S, Mclendon P, Campbell M, Alway S, Efymow B, Gracia C. Oocyte cryopreservation in a patient with sickle cell disease prior to hematopoietic stem cell transplantation: first report. J Assist Reprod Genet. 2012 Mar;29(3):265-9. doi: 10.1007/s10815-011-9698-2. Epub 2012 Jan 5. PMID 22219083